CLINICAL TRIAL: NCT03012282
Title: Evaluation of CT Perfusion Parameters as a Potential Biomarker for Treatment Response in Pancreatic Cancer
Brief Title: CT Perfusion Images in Assessing Treatment Response in Patients With Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination due to slow accrual
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9625; NCI-2016-01780 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9625 (Other: Fred Hutch/University of Washington Cancer Consortium); RG3017007 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (CT perfusion sequence) (Experimental): Patients undergo CT perfusion sequence during the first 40 seconds of the baseline standard of care CT scan and during follow-up CT scans at 2 and possibly 4 months after chemotherapy, at 4-6 weeks after radiation therapy, or prior to definitive surgery.
  Interventions: Diagnostic Test: Computed Tomography Perfusion Imaging

INTERVENTIONS:
Diagnostic Test: Computed Tomography Perfusion Imaging — Undergo CT perfusion sequence

SUMMARY:
This pilot clinical trial studies how well computed tomography (CT) perfusion images work in assessing treatment response in patients with pancreatic cancer. Analyzing specific measurements on the CT perfusion images may help doctors better determine how a tumor responds to chemotherapy and/or radiation therapy and may help guide treatment for patients with pancreatic cancer.

DETAILED DESCRIPTION:
OUTLINE:

Patients undergo CT perfusion sequence during the first 40 seconds of the baseline standard of care CT scan and during follow-up CT scans at 2 and possibly 4 months after chemotherapy, at 4-6 weeks after radiation therapy, or prior to definitive surgery.

After completion of the study, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* A diagnosis of pancreatic ductal adenocarcinoma

Exclusion Criteria:

* Patients unable to provide informed consent
* Women who are pregnant or intending to become pregnant during the study
* Patients with body mass index greater than 40 kg/m^2
* History of severe allergic-like reaction to iodinated contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Correlation between pre-treatment computed tomography (CT) tumor perfusion parameters and percentage of patients who achieve curative (R0) surgical resection after neoadjuvant chemotherapy | Up to 4 years
  Assessed using logistic regression. Receiver operating characteristic (ROC) curve analysis will be used to examine the sensitivity and specificity of different thresholds for each parameter.
Correlation between pre-treatment CT tumor perfusion parameters and tumor response after treatment | Up to 1 year
  Will be defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Assessed using logistic regression. ROC curve analysis will be used to examine the sensitivity and specificity of different thresholds for each parameter. If multiple perfusion parameters are found to be predictive of response, a multivariate logistic regression model will be constructed with these variables. ROC analysis will also be used to summary the predictive performance of the multivariate model.
Correlation of pre-treatment CT tumor perfusion parameters with overall survival | At 1 year
  Assessed using Cox regression models. Multivariate Cox models will be constructed if multiple parameters are found to be predictive of survival.
Correlation of pre-treatment CT tumor perfusion parameters with overall survival | At 2 years
  Assessed using Cox regression models. Multivariate Cox models will be constructed if multiple parameters are found to be predictive of survival.
Correlation of pre-treatment CT tumor perfusion parameters with progression free survival | At 1 year
  Assessed using Cox regression models. Multivariate Cox models will be constructed if multiple parameters are found to be predictive of survival.
Correlation of pre-treatment CT tumor perfusion parameters with progression free survival | At 2 years
  Assessed using Cox regression models. Multivariate Cox models will be constructed if multiple parameters are found to be predictive of survival.
Change in computed tomography (CT) tumor perfusion parameters (time to peak concentration) | Baseline to post-treatment (up to approximately one year)
  The change in each CT tumor perfusion parameter between the pre-treatment scan and the post-treatment scan where response is assessed will be calculated. These changes will be compared between the responders and non-responders using the t-test or Mann-Whitney test.
Change in CT tumor perfusion parameter (blood flow) | Baseline to post-treatment (up to approximately one year)
  The change in each CT tumor perfusion parameter between the pre-treatment scan and the post-treatment scan where response is assessed will be calculated. These changes will be compared between the responders and non-responders using the t-test or Mann-Whitney test.
Change in CT tumor perfusion parameter (blood volume) | Baseline to post-treatment (up to approximately one year)
  The change in each CT tumor perfusion parameter between the pre-treatment scan and the post-treatment scan where response is assessed will be calculated. These changes will be compared between the responders and non-responders using the t-test or Mann-Whitney test.
Change in CT tumor perfusion parameter (Ktrans) | Baseline to post-treatment (up to approximately one year)
  The change in each CT tumor perfusion parameter between the pre-treatment scan and the post-treatment scan where response is assessed will be calculated. These changes will be compared between the responders and non-responders using the t-test or Mann-Whitney test.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan O'Malley, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No